CLINICAL TRIAL: NCT04248517
Title: Using mHealth to Optimize Pharmacotherapy Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Northwell Health, Early Treatment Program at Lenox Hill (Unknown); The Institute for Family Health Center for Counseling at Walton (Unknown); New York State Psychiatric Institute, Washington Heights Community Service (Unknown); BestSelf Behavioral Health (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Scott Stroup, Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7900; P50MH115843 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; First-Episode Psychosis
Keywords: mHealth; Schizophrenia; EMA
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Prospective cohort with comparison group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth intervention group (Experimental): participants in the mHealth Group will download the app on to their smartphone and complete ecological momentary assessments on 3 consecutive weekdays every 2 weeks for 6 months.
  Interventions: Other: mHealth Intervention
- Treatment as Usual group (No Intervention): participants will undergo their routine treatment.

INTERVENTIONS:
Other: mHealth Intervention — Participants will download the app onto their smartphone and complete ecological momentary assessements
  Arms: mHealth intervention group

SUMMARY:
This project will use a smartphone technology to improve medication prescribing for individuals with FEP. We will collect real-time symptom and functioning data via smartphones to provide prescribers and other clinical team members with clinically relevant and time-sensitive information that will inform and promote shared decision making (SDM) and personalized interventions. The result will be a time-sensitive, data-driven, collaborative process to optimize medication regimens in order to maximize benefits, minimize harms, and promote adherence.

DETAILED DESCRIPTION:
Comprehensive early treatment of individuals experiencing schizophrenia has the potential to alter the course of illness and improve long-term outcomes. Psychotropic medications are a critical component of early treatment strategies. First-episode psychosis (FEP) is a critical time to optimize prescribing but evidence suggests that prescribing for this population is suboptimal.

A contributing factor to these difficulties is thought to be the lack of accurate information about the effects of medications on symptoms, their side effects, as well as their behavioral, cognitive, and emotional correlates. At medication management appointments, prescribers typically rely on patients' recollection of how they were doing over periods of weeks. Such retrospective assessments are problematic as they are vulnerable to the influence of memory difficulties, cognitive biases including recency effects and frequency illusions, and reframing. Recent advances in smartphone technologies (mobile Health; mHealth) may help to overcome many of the limitations of retrospective assessments.

This pilot study will be a collaboration with OnTrackNY, an innovative coordinated specialty care (CSC) program for individuals aged 16-30 who are experiencing FEP. OnTrackNY originated as part of the NIMH Recovery After an Initial Schizophrenia Episode (RAISE) Implementation and Evaluatoin Study. The initial phase of this project will use input from stakeholders including patients, front-line providers, clinical leaders, and members of the research team to adapt and refine the mHealth intervention to improve feasibility and clinical utility. A pilot study at 3 OnTrackNY sites will then examine its feasibility and effectiveness by comparing the management and outcomes of 60 patients randomly assigned to the mHealth application or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female OnTrackNY participants, ages 16 to 30, of any race/ethnicity
* Able and willing to give informed consent and participate in the intervention
* Participating in OnTrackNY for less than 1 year because this group may be more in need of medication adjustments and will be less likely to graduate from the program before 6 months of participation.

Exclusion Criteria:

* Suicidal at baseline with C-SSRS score 4 or 5.
* PANSS baseline score of 5 (moderately severe) or greater on the Conceptual Disorganization item (P2)

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
change of Treatment Satisfaction Questionnaire for Medication (TQSM) from baseline to 6 months | baseline to 6 months
  The TSQM assesses client satisfaction with medication. It comprises 14 items across four domains focusing on effectiveness (3 items), side effects (5 items), convenience (3 items), and global satisfaction (3 items) of the medication over the previous 2-3 weeks, or since the patient's last use. With the exception of item 4 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied).The 7-item scales had a non-neutral midpoint, such that there were more positive response options than negative response options, to allow for precise information to be obtained at the upper end of the score distribution. Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100. Item 4 was not included for scoring. If an item score is missing and half of the items in the domain are complete, domain scores may be imputed from the person-specific mean score of completed items.
change of Client Satisfaction Questionnaire (CSQ-8) from baseline to 6 months | baseline to 6 months
  8-item easily scored and administered measurement that is designed to measure client satisfaction with services. The overall score is produced by summing all item responses. Scores range from 8 to 32, with higher values indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stroup, MD, MPH, Principal Investigator — New York State Psychiatric Institute
Locations (4):
- United States (4):
  - Bestself Behavioral Health, Inc., Buffalo, New York
  - Washington Heights Community Service, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Institute for Family Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories including the National Database for Clinical Trials related to Mental Illness (NDCT). Data will include baseline demographic data, and baseline and post raw data derived from functioning and symptom measures.
Supporting Information: Study Protocol
Time Frame: A list of all data expected to be collected in the project will be submitted within 6 months of award. Subsequently, descriptive and raw data will be submitted on a semi-annual basis. Unpublished de-identified data will be submitted prior to study completion and will be shared within one year after project completion, or when the data are published, whichever is earlier.
Access Criteria: Data in NIH repositories may be accessed through the NIH Data Access Committee which reviews data access and submission requests.

REFERENCES:
- [Derived] Stefancic A, Rogers RT, Styke S, Xu X, Buchsbaum R, Nossel I, Cabassa LJ, Stroup TS, Kimhy D. Development of the First Episode Digital Monitoring mHealth Intervention for People With Early Psychosis: Qualitative Interview Study With Clinicians. JMIR Ment Health. 2022 Nov 4;9(11):e41482. doi: 10.2196/41482. PMID 36331539